CLINICAL TRIAL: NCT02857751
Title: Evaluation of Health Outcomes Following the NMCSD Surf Therapy Program
Brief Title: Evaluation of Outcomes Following Surf Therapy
Status: Completed | Type: Observational
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: Naval Health Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kristen Walter, Clinical Research Psychologist, United States Naval Medical Center, San Diego
Other Study IDs: NMCSD.2016.0032
Record Dates: First submitted 2016-07-13; First posted 2016-08-05 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Depression; Posttraumatic Stress Disorder
Keywords: depression; PTSD; anxiety; surf therapy
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Surf therapy cohort 1: The first cohort of participants to enroll in the study (i.e., participants in the first 6-week program)
  Interventions: Behavioral: Surf therapy
- Surf therapy cohort 2: The second cohort of participants to enroll in the study (i.e., participants in the second 6-week program)
  Interventions: Behavioral: Surf therapy
- Surf therapy cohort 3: The third cohort of participants to enroll in the study (i.e., participants in the third 6-week program)
  Interventions: Behavioral: Surf therapy
- Surf therapy cohort 4: The fourth cohort of participants to enroll in the study (i.e., participants in the fourth 6-week program)
  Interventions: Behavioral: Surf therapy
- Surf therapy cohort 5: The fifth cohort of participants to enroll in the study (i.e., participants in the fifth 6-week program)
  Interventions: Behavioral: Surf therapy

INTERVENTIONS:
Behavioral: Surf therapy — The NMCSD surf therapy program is approximately 6 weeks in duration. Each surf therapy session lasts 2-3 hours and occurs in a group setting that can accommodate up to 20 service members per session. Each service member is paired with a surf instructor who works with him or her each week for the 6-week session. Goals are individually-tailored to the service member (based on participant's level of comfort in the water, experience with surfing, etc.) and can incorporate both physical and psychological objectives.

SUMMARY:
The current study evaluates psychological and physical health outcomes for active-duty service members following participation in an established surf therapy program. Participants complete assessments before and after the surf therapy program, as well as brief assessments before and after each surf therapy session.

DETAILED DESCRIPTION:
The proposed study would evaluate whether an existing surf therapy program that is part of the Wounded, Ill, and Injured (WII) Wellness Program at Naval Medical Center San Diego (NMCSD), significantly reduces both psychological symptoms (e.g., PTSD, depression, anxiety, negative affect, lack of positive affect) and physical symptoms (e.g., pain, sleep) among active-duty service members. Psychological and physical symptoms will be assessed before beginning the surf program and at program completion. In addition, brief assessments of mood and symptoms will be completed before and after each individual surf therapy session.

ELIGIBILITY:
Inclusion Criteria:

* Active-duty military service members seeking surf therapy at NMCSD and have been medically cleared to participate
* Diagnosis of either a psychological (e.g., PTSD, depression) or physical (e.g., amputated limb; traumatic brain injury) condition that served as a reason for referral

Exclusion Criteria:

* Service members who cannot receive medical clearance to participate in the NMCSD surf therapy program
* Service members who have previously participated in the NMCSD surf therapy program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample will consist of up to 75 active-duty service members (male or female) who are seeking surf therapy through the WII Wellness Program at NMCSD. As the study is being implemented into standard care, the current study is designed to have broad eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-8) | From pre- to post-program (e.g., approximately 6-8 weeks)
  Self-reported depression symptoms

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | From pre- to post-program (e.g., approximately 6-8 weeks)
  Report of satisfaction with the surf therapy program

CONTACTS AND LOCATIONS:
Overall Officials: Betty Michalewicz-Kragh, M.S., Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Walter, K. H., Otis, N. P., Ray, T. N., Powell, A. L., Glassman, L. H., Michalewicz-Kragh, B., & Thomsen, C. J. (2019). Breaking the Surface: Psychological Outcomes among U.S. active duty service members following a surf therapy program. Psychology of Sport and Exercise. doi: 10.1016/j.psychsport.2019.101551
- [Result] Otis, N. P., Walter, K. H., Glassman, L. H., Ray, T. N., Michalewicz-Kragh, B., & Thomsen, C. J. (2020). Effects of PTSD and MDD comorbidity on psychological changes during surf therapy sessions for active duty service members. Special Issue of Global Journal of Community Psychology and Practice on Surf Therapy. https://www.gjcpp.org/en/article.php?issue=36&article=210
- [Result] Glassman LH, Otis NP, Michalewicz-Kragh B, Walter KH. Gender Differences in Psychological Outcomes Following Surf Therapy Sessions among U.S. Service Members. Int J Environ Res Public Health. 2021 Apr 27;18(9):4634. doi: 10.3390/ijerph18094634. PMID 33925447